CLINICAL TRIAL: NCT04871074
Title: SV2A PET Imaging in Alzheimer's Disease
Brief Title: The Synapse Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-1283; A534255 (Other: UW Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison); Protocol Version 3/7/2024 (Other: UW Madison); R01AG062285 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cognitively Impaired plus Cognitive Unimpaired Participants (Experimental): Participants include both cognitively impaired and unimpaired populations to populate a single model to examine variables within the group as a whole.
  * Cognitively impaired participants have abnormal cognitive status of MCI or dementia as judged by consensus or expert review using National Institute of Aging and Alzheimer's Association (NIA-AA) 2018 criteria.
  * Cognitively unimpaired participants: results of most recent testing with the source cohort indicate the participant is cognitively unimpaired as judged by consensus or expert review.
  Interventions: Drug: UCB-J; Device: MRI Scan; Device: PET Scan

INTERVENTIONS:
Drug: UCB-J — PET imaging with UCB-J
Device: MRI Scan — MRI exams will be performed using a 3T MRI scanner, scan duration is typically 60 minutes
  Other Names: Magnetic Resonance Imaging
Device: PET Scan — PET imaging may be collected using either a PET scanner or a PET/Computed Tomography (CT) scanner, a PET scan will be initiated with the injection of radiotracer
  Other Names: Positron Emission Tomography

SUMMARY:
The overarching goal of this project is to use [C-11]UCB-J to obtain spatial information on neuronal synapse abundance and inform Alzheimer's disease (AD) progression. The investigators propose to collect longitudinal amyloid, tau, and Synaptic vesicle glycoprotein 2A (SV2A) positron emission tomography (PET) in participants in the Wisconsin Alzheimer's Disease Research Center (ADRC) and Wisconsin Registry for Alzheimer's Prevention (WRAP) across the clinical stages of AD, including cognitively unimpaired biomarker negative, unimpaired biomarker positive, mild cognitive impairment (MCI), and dementia due to AD.

DETAILED DESCRIPTION:
Synaptic loss is a major feature of symptomatic AD. Conversely, abundance of synapses may confer resilience to cognitive decline in the presence of AD pathology. The pathology-defining features of AD are amyloid plaques and neurofibrillary tangles and their presence and distribution can be spatially estimated in-vivo with amyloid and tau PET. Although these biomarkers can inform on the degree and location of pathology, they do not provide an indicator of their effect on collocated or extended in-network neural damage including synaptic density.

SV2A is expressed ubiquitously in synapses and the capability of assessing SV2A in vivo may provide a direct indicator of synaptic health. Such information would be of high importance for staging the level of synaptic loss or conversely synaptic abundance in the AD continuum and may potentially improve prognostic precision. The PET radioligand [C-11]UCB-J is a marker of SV2A.

The overarching goal of this project is to use [C-11]UCB-J to obtain spatial information on neuronal synapse abundance and inform upon disease progression. The investigators propose to collect longitudinal amyloid, tau, and SV2A PET in participants in the Wisconsin ADRC and WRAP across the clinical stages of AD, including cognitively unimpaired biomarker negative, unimpaired biomarker positive, MCI, and dementia due to AD.

* Specific Aim 1). Determine the extent to which [C-11]UCB-J provides unique information from MRI regarding neurodegeneration. Approach: The investigators will recruit N=60 cognitively unimpaired participants, N=30 MCI participants, and N=30 participants with AD dementia to undergo PET imaging with [C-11]UCB-J. MRI will include anatomic and diffusion connectivity MRI. When available, ancillary cerebrospinal fluid (CSF) indicators of neurodegeneration and synapse function will be examined for relationships with UCB-J.
* Specific Aim 2). Determine the rate of synapse loss as reflected by [C-11]UCB-J signal across all participants. Rationale: Trajectories of synaptic loss are unknown in vivo. Approach: The investigators will determine the longitudinal trajectories of regional synapse loss that are observed over time among participants who undergo repeat [C-11]UCB-J (separated by two years, same participants scanned for Aim 1). The investigators will also examine trajectories by amyloid and tau load. Quantifying longitudinal synaptic loss is expected to eventually facilitate the identification of individuals who are progressing to dementia, as well as inform upon changes that are normal for age.
* Specific Aim 3). Determine the extent to which [C-11]UCB-J associates with cognitive decline. Rationale: The investigators expect that lower baseline SV2A density and longitudinal decline in SV2A density in the medial temporal lobe will be associated with faster progression of cognitive decline. The investigators will also test the extent to which harboring multiple pathologies (↑amyloid, ↑tau, and ↓SV2A density) contributes to cognitive decline. Approach: The investigators will examine core indices of cognitive status and continuous measures of cognitive function from the source cohorts and utilize mixed effects models to ascertain the effect of UCB-J amyloid and tau on cognition.
* Specific Aim 4). Determine factors which impact synapse loss. Rationale: Several risk factors for cognitive decline and dementia have been identified including potentially modifiable factors such as insulin resistance and vascular risk factors. Approach: The investigators will determine cross-sectional and longitudinal trajectories of regional synapse loss in relation to risk factors for cognitive decline and dementia. In order to determine insulin resistance, the investigators will perform blood draw and assess fasting glucose and insulin values to determine the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). The impact of potentially modifiable risk factors on synapse loss in vivo is currently unknown. This aim will address this gap in knowledge, results which may translate to strategies for reducing dementia risk.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively unimpaired adults-

  * Aged 55 - 89
  * Normal cognition (results of most recent testing with the source cohort indicate the participant is cognitively unimpaired as judged by consensus or expert review)
  * In good general health with no conditions/medications affecting cognition or imaging
  * Willing to undergo [C-11]UCB-J, [C-11]PiB, and [F-18]MK6240 PET scans
  * An adequate MRI exam within 12 months prior to baseline. An MRI will be performed if not already available.
* Mild dementia and amnestic Mild Cognitive Impairment-

  * Aged 50 years or older
  * Abnormal cognitive status of MCI or dementia as judged by consensus or expert review using NIA-AA 2018 criteria
  * MCI's must be affected in the memory domain but may also have other affected domains
  * Willing to undergo [C-11]UCB-J, [C-11]PiB, and [F-18]MK6240 PET scans
  * An adequate MRI exam within 12 months prior to baseline. This MRI exam will come from ADRC/WRAP studies. Clinical MRI's (ones obtained outside of the research program) will not be adequate. An MRI will be performed if not already available from within the research program.

Exclusion Criteria:

* For women, pregnant, lactating or breastfeeding, or intention to become pregnant
* Evidence of unstable or untreated clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Stable, treated chronic medical conditions like hypertension, hypercholesterolemia, diabetes mellitus, non-metastatic dermatologic or prostatic cancer, etc. are acceptable as long as they do not, in the study investigator's opinion, contribute to cognitive dysfunction or limit participation in study procedures.
* Any illness or other consideration that makes it unlikely that the subject will be able to complete the 24-month study.
* Current or prior history (within past 5 years) of significant alcohol or substance abuse as determined by the investigator.
* Psychiatric disorders that may interfere with the study including current major Axis I DSM-V disorders including but not limited to severe Major depression, current or history of bipolar I disorder, or schizophrenia.
* Current use of the anti-seizure medication Levetiracetam, also known as Keppra, Spritam or Roweepra
* MRI exclusion criteria include findings from previous MRI's within the ADRC/WRAP research program that may be responsible for neurologic status of the subject such as evidence of cerebrovascular disease with multiple infarcts, infectious disease, space-occupying lesion, normal pressure hydrocephalus, CNS trauma, or any other structural abnormality that may impact cognition or image analysis, as judged by the investigator.
* MRI-incompatible implants or devices such as certain cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI that prevents completion of MRI protocol.
* Lack of decisional capacity at the time of informed consent
* Lumbar puncture exclusion criteria include: previous lumbar spine surgery, currently taking blood-thinning anti-platelet medications, taking immunosuppressive medications, currently being treated or were recently treated for an infection or virus within the last 2 to 3 months.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bendlin, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The intent of the study was observational, to characterize synaptic density across disease stages, the groups shown in the Baseline Characteristic Section are non-randomized subgroups within a single study arm.
Period: Overall Study
Arm/Group | Cognitively Impaired Plus Cognitive Unimpaired Participants
Started | 100
Cognitively Unimpaired Subgroup | 65
Cognitively Impaired Subgroup | 35
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The intent of the study was observational, to characterize synaptic density across disease stages, the groups shown in the Baseline Characteristic Section are non-randomized subgroups within a single study arm.
Groups:
- Cognitively Unimpaired: Results of most recent testing with the source cohort indicate the participant is cognitively unimpaired as judged by consensus or expert review.
- Cognitively Impaired: Abnormal cognitive status of MCI and Dementia as judged by consensus or expert review using National Institute of Aging and Alzheimer's Association (NIA-AA) 2018 criteria.
- Total: Total of all reporting groups
Arm/Group | Cognitively Unimpaired | Cognitively Impaired | Total
Number analyzed (Participants) | 65 | 35 | 100
Age, Continuous [Mean (Full Range); unit: years] | 68.9 [56.3 to 89.8] | 75.2 [63.0 to 86.4] | 71.1 [56.3 to 89.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 11 | 56
  Male | 20 | 24 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 65 | 35 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 54 | 31 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 65 | 35 | 100
Cognitive Impairment [Count of Participants; unit: Participants] — Population: Not applicable to this group
  Participants
    number analyzed (Participants) | 0 | 35 | 35
    Mild Cognitive Impairment | 0 | 22 | 22
    Mild Dementia | 0 | 13 | 13

OUTCOME MEASURES:

1. Primary Outcome: ROC AUCs (MCI/AD vs Cognitively Unimpaired (CU)) for Medial Temporal Lobe (MTL) UCB-J Distribution Volume Ratio (DVR) and Hippocampal Volume
Description: DeLong's method will test whether the MTL UCB-J receiver-operator characteristic (ROC) area under the curve (AUC) has better mild cognitive impairment/probable AD dementia (MCI/AD) prediction accuracy than the hippocampal volume ROC AUC. ROC AUC is a measure of the correctness of group (where group is MCI/AD and cognitively unimpaired) classification using a continuous predictor, in this case, the medial temporal lobe UCB-J uptake (11C-UCB-J is a PET tracer for imaging the synaptic vesicle glycoprotein 2A in the human brain. It is considered a measure of synaptic density). This ROC AUC was compared to that of the comparator continuous predictor, hippocampal volume.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Medial Temporal Lobe UCB-J: Synaptic density in the Medial Temporal Lobe across all participants
- Hippocampal Volume: Hippocampal volume across all participants
Arm/Group | Medial Temporal Lobe UCB-J | Hippocampal Volume
Number analyzed (Participants) | 100 | 100
probability | 0.79 [0.68 to 0.89] | 0.81 [0.71 to 0.91]
Statistical Analysis 1: Comparison: Medial Temporal Lobe UCB-J vs Hippocampal Volume; Test type: Superiority; p = .74, DeLong's Test

2. Primary Outcome: ROC AUCs (MCI/AD vs CU) for MTL UCB-J and Hippocampal Cingulum Neurite Density Index
Description: DeLong's method will test whether the MTL UCB-J ROC AUC has better MCI/AD prediction accuracy than the hippocampal cingulum neurite density index ROC AUC. ROC AUC is a measure of the correctness of group (where group is MCI/AD and cognitively unimpaired) classification using a continuous predictor, in this case, the medial temporal lobe UCB-J uptake (11C-UCB-J is a PET tracer for imaging the synaptic vesicle glycoprotein 2A in the human brain. It is considered a measure of synaptic density). This ROC AUC was compared to that of the comparator continuous predictor, hippocampal cingulum neurite density index.
Time Frame: Baseline
Population: Usable data on 79 participants (due to processing)
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Hippocampal Cingulum NDI: Neurite density index (NDI) in the Hippocampal Cingulum across all participants
Arm/Group | Medial Temporal Lobe UCB-J | Hippocampal Cingulum NDI
Number analyzed (Participants) | 79 | 79
probability | 0.82 [0.71 to 0.93] | 0.79 [0.69 to 0.89]
Statistical Analysis 1: Comparison: Medial Temporal Lobe UCB-J vs Hippocampal Cingulum NDI; Test type: Superiority; p = .66, DeLong's Test

3. Primary Outcome: Annual Rate of Change in UCB-J DVR
Description: Linear mixed effects regression will model UCB-J distribution volume ratio (DVR) as a function of time since baseline. 11C-UCB-J is a PET tracer for imaging the synaptic vesicle glycoprotein 2A in the human brain. It is considered a measure of synaptic density. Participants' synaptic density was examined as a change per year. A positive number would mean an increase in synaptic density, a negative number means a decrease.
Time Frame: Baseline and 2 years
Population: N = 25 contributing to the time estimate
Measure: Number (95% Confidence Interval); unit: distribution volume ratio per year
Groups:
- All Participants: Cognitively unimpaired and cognitively impaired participants
Arm/Group | All Participants
Number analyzed (Participants) | 100
distribution volume ratio per year | -.01 [-.02 to 0]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = .135, Mixed Models Analysis; Linear mixed effects model, fixed effects coefficient test with a Wald test

4. Primary Outcome: Baseline Diagnosis Group Differences in Annual Rate of Change in UCB-J DVR
Description: Baseline diagnosis (CU vs MCI/probable AD dementia) group differences in rate of UCB-J DVR change will be estimated via group x time interaction term in a linear mixed effects model. Participants' synaptic density was examined as a change per year. The difference in the rate of change in the two groups was estimated. A negative number means that impaired participants decreased in synaptic density more quickly and a positive number would mean that the impaired participants decreased less quickly.
Time Frame: baseline and 2 years
Population: While 100 participants were enrolled in the study and entered into the model, 25 participants were measured at follow up and contributed to the time estimate; among those 25, 7 cognitively impaired and 18 unimpaired.
Measure: Number (95% Confidence Interval); unit: distribution volume ratio per year
Arm/Group | Cognitively Unimpaired | Cognitively Impaired
Number analyzed (Participants) | 65 | 35
distribution volume ratio per year | 0 [-.02 to .01] | -.02 [-.04 to 0]

5. Primary Outcome: Amyloid Positivity Status Differences in Annual Rate of Change in UCB-J DVR
Description: Amyloid positivity status differences in rate of UCB-J DVR change will be estimated via group x time interaction term in a linear mixed effects model. Amyloid positivity status will be determined from amyloid PET. Participants' synaptic density was examined in a change per year. The difference in the rate of change in the two groups was estimated. A negative number means that amyloid positive participants decreased in synaptic density more quickly and a positive number would mean that the amyloid positive participants decreased less quickly.
Time Frame: baseline and 2 years
Population: 90 people contributed to the overall model, 24 participants contributed to the time estimate; 3 Amyloid positive, 21 Amyloid negative, centiloid values for amyloid scans unavailable for 10 participants (unable to process)
Measure: Number (95% Confidence Interval); unit: distribution volume ratio per year
Groups:
- Amyloid Positive: Amyloid Positive
- Amyloid Negative: Amyloid Negative
Arm/Group | Amyloid Positive | Amyloid Negative
Number analyzed (Participants) | 43 | 47
distribution volume ratio per year | -.02 [-.05 to .01] | -.01 [-.02 to 0]

6. Primary Outcome: Tau Positivity Status Differences in Annual Rate of Change in UCB-J DVR
Description: Tau positivity status differences in rate of UCB-J DVR change will be estimated via group x time interaction term in a linear mixed effects model. Tau positivity status will be determined from tau PET. Participants' synaptic density was examined as a change per year. The difference in the rate of change in the two groups was estimated. A negative number means that tau positive participants decreased in synaptic density more quickly and a positive number would mean that the tau positive participants decreased less quickly.
Time Frame: baseline and 2 years
Population: While 94 participants were included in the model, 24 participants contributed to the time estimate; 1 Tau positive, 23 Tau negative, tau status unavailable for 6 participants, no data available for Tau scan.
Measure: Number (95% Confidence Interval); unit: distribution volume ratio per year
Groups:
- Tau Positive: Tau Positive
- Tau Negative: Tau Negative
Arm/Group | Tau Positive | Tau Negative
Number analyzed (Participants) | 38 | 56
distribution volume ratio per year | -.02 [-.08 to .04] | -.01 [-.02 to 0]

7. Primary Outcome: MTL UCB-J DVR Baseline Differences in a Cognitive Performance Age Slope in Non-demented Participants
Description: Linear mixed effects will be used to model cognitively unimpaired participants' memory performance as a function of their age and synaptic density. Specifically, investigators will test whether those with higher synaptic density had less deterioration over time. Memory performance will be assessed using Rey Auditory Verbal Learning Test Delayed Recall. An interaction was tested, and a negative number means that those with higher synaptic density decreased faster over time, and a positive number means that they decreased slower over time.
Time Frame: baseline and 2 years
Measure: Number (95% Confidence Interval); unit: diff in rate of change AVLT per year
Groups:
- Cognitively Unimpaired: Cognitively unimpaired participants
Arm/Group | Cognitively Unimpaired
Number analyzed (Participants) | 65
diff in rate of change AVLT per year | -.05 [-.17 to .07]
Statistical Analysis 1: Comparison: Cognitively Unimpaired; Test type: Superiority; p = .39, Mixed Models Analysis; Fixed effects estimate, Wald test

8. Secondary Outcome: Difference Between ROC AUCs (MCI/AD vs CU) for Medial Temporal Lobe (MTL) UCB-J Distribution Volume Ratio (DVR) and Cerebrospinal Fluid (CSF) Neurofilament Light Chain Protein (NfL)
Description: DeLong's method will test whether the MTL UCB-J ROC AUC has better mild cognitive impairment/probable AD dementia (MCI/AD) prediction accuracy than the CSF NfL ROC AUC.
Time Frame: baseline
Reporting Status: Not Posted, anticipated posting 2026-01

9. Secondary Outcome: Difference Between ROC AUCs (MCI/AD vs CU) for MTL UCB-J DVR and Cerebrospinal Fluid (CSF) T-tau
Description: DeLong's method will test whether the MTL UCB-J ROC AUC has better MCI/AD prediction accuracy than the CSF T-tau ROC AUC.
Time Frame: baseline
Reporting Status: Not Posted, anticipated posting 2026-01

10. Secondary Outcome: Difference Between ROC AUCs (MCI/AD vs CU) for MTL UCB-J and CSF Neurogranin
Description: DeLong's method will test whether the MTL UCB-J ROC AUC has better MCI/AD prediction accuracy than the CSF neurogranin ROC AUC.
Time Frame: baseline
Reporting Status: Not Posted, anticipated posting 2026-01

11. Secondary Outcome: Sex Differences in Annual Rate of Change in UCB-J DVR
Description: Sex differences in rate of UCB-J DVR change will be estimated via group x time interaction term in a linear mixed effects model.
Time Frame: baseline and 2 years
Reporting Status: Not Posted, anticipated posting 2026-01

12. Secondary Outcome: Age Differences in Annual Rate of Change in UCB-J DVR
Description: Age differences in rate of UCB-J DVR change will be estimated in a linear mixed effects model.
Time Frame: baseline and 2 years
Reporting Status: Not Posted, anticipated posting 2026-01

13. Secondary Outcome: APOE4 Allele Status Differences in Annual Rate of Change in UCB-J DVR
Description: APOE4 allele status differences in rate of UCB-J DVR change will be estimated via group x time interaction term in a linear mixed effects model.
Time Frame: baseline and 2 years
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: data collected during study contact, up to 2 years on study
Groups:
- Cognitively Impaired: Abnormal cognitive status of MCI or dementia as judged by consensus or expert review using National Institute of Aging and Alzheimer's Association (NIA-AA) 2018 criteria.
Arm/Group | Cognitively Unimpaired | Cognitively Impaired
All-Cause Mortality (participants affected / at risk) | 0/65 | 3/35
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/35
Other Adverse Events (participants affected / at risk) | 21/65 | 5/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitively Unimpaired (N=65) | Cognitively Impaired (N=35)
Transient Visual Disturbance (Eye disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1)
Brain Fog (Psychiatric disorders) | 1 (1) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scab on Back of Head (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (10) | 1 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
"Fizzies" in both legs (Nervous system disorders) | 1 (1) | 0 (0)
Presyncopy (Nervous system disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Coolness (General disorders) | 1 (1) | 0 (0) — "coolness" energy travelling up both sides of face up to temples
Confusion and Headache (Psychiatric disorders) | 1 (1) | 0 (0) — disoriented on drive home and mild headache
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Anosmia (General disorders) | 1 (1) | 0 (0) — smelled something odd

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04871074/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04871074/ICF_001.pdf